CLINICAL TRIAL: NCT06909877
Title: An Open-label, Multinational, Multicenter, Single-arm Phase Ⅰb/Ⅱ Study to Evaluate Efficacy and Safety of Oral HH2853, a Selective EZH1/2 Inhibitor, in Patients With Relapsed/Refractory Peripheral T-cell Lymphoma
Brief Title: Study to Evaluate Efficacy and Safety of HH2853 in Relapsed/Refractory Peripheral T-cell Lymphoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Haihe Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HH2853-G202
Record Dates: First submitted 2025-03-20; First posted 2025-04-04 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Relapsed/Refractory Peripheral T-Cell Lymphoma (R/R PTCL)
Keywords: Relapsed/Refractory; Peripheral T-cell Lymphoma
MeSH Terms: conditions — Recurrence; Lymphoma, T-Cell, Peripheral

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose escalation and expansion study of HH2853 (Experimental): To determine the RP2D of HH2853 in PTCL patients.
  Interventions: Drug: HH2853 Tablets

INTERVENTIONS:
Drug: HH2853 Tablets — 25mg, 100mg and 200 mg BID oral administration
  Other Names: HH2853

SUMMARY:
This study is a an open-label, multinational, multicenter, single-arm Phase Ⅰb/Ⅱ Study to Evaluate Efficacy and Safety of Oral HH2853 in Patients with Relapsed/Refractory Peripheral T-cell Lymphoma.

DETAILED DESCRIPTION:
This study includes Phase Ib and Phase II. In the Phase Ib, patients with R/R NHL (dose escalation) or R/R PTCL (dose expansion) who have received at least 1 line of prior systematic treatment and meet the inclusion/exclusion criteria in the protocol will be enrolled. Safety run-in study (Japan only): The objective of the safety run-in study in Japan is to evaluate the safety, tolerability, and PK profile of HH2853 in Japanese patients. The primary objective of the Phase Ib study is to determine the RP2D of HH2853 in PTCL patients. The secondary objectives are to evaluate the safety, preliminary efficacy and characterize the pharmacokinetic profile of HH2853 in R/R PTCL patients. A "3+3" design will be used in the dose escalation part with a starting dose of 400 mg BID. Based on the safety, efficacy and PK/PD data and HH2853-G101 data, 1-2 dose levels could be expanded, 10-15 R/R PTCL patients for each dose level. Approximately 21-48 patients will be enrolled in total.

In the Phase II (multi-national): patients with R/R PTCL who have received at least one prior systemic combination chemotherapy and at least one new drug therapy and meet the inclusion/exclusion criteria in the protocol will be enrolled. The Phase II study will be started once the RP2D is determined. The Phase II study is a single-arm study and will be enrolled in approximately 66 efficacy-evaluable R/R PTCL patients who had received at least one prior systemic combination chemotherapy and at least one new drug therapy. The primary objective of the Phase II study is to evaluate the efficacy of HH2853 of R/R PTCL patients who have received at least one prior systemic combination chemotherapy and at least one new drug therapy (ORR, BIRC evaluation); The secondary objectives will be continued to further evaluate the efficacy, safety, tolerability and PK characteristics of HH2853 of R/R PTCL patients who have received at least 1 line of prior systemic therapy.

ELIGIBILITY:
Inclusion Criteria:

* main inclusion:

  1. Tumor types and prior antitumor therapy: Phase Ib:Dose Escalation: All enrolled patients must have histologically confirmed diagnosis NHL who have received at least one line of prior systematic treatment (and ≤ 5 lines) and relapses or refractory. Phase Ib dose expansion part: All enrolled patients must have histologically confirmed diagnosis of PTCL, including subtypes: PTCL-NOS, AITL, ALK + ALCL, ALK-ALCL, NKTCL, enteropathy associated T-cell lymphoma (EATL), monomorphic epitheliotropic internal T-cell lymphoma (MEITL), Hepatosplenic T-cell lymphoma (HSTCL), follicular T-cell lymphoma (FTCL), Nodal peripheral T-cell lymphoma with TFH phenotype (Nodal PTCL-TFH) and other invasive T-cell sources NHL at the investigator and sponsor's discretion (except highly invasive). All enrolled patients had relapsed or refractory diseases after receiving 1-line systematic treatment (≤ 3 lines). Phase II: All enrolled patients must have histologically confirmed diagnosis of PTCL, including subtypes: PTCL-NOS, AITL, ALK+ALCL, ALK-ALCL, NKTCL, EATL, MEITL, HSTCL, FTCL, Nodal PTCL-TFH et al. Patients must have histologically confirmed diagnosis of R/R PTCL who have received at least one line of prior systematic combination chemotherapy and at least one new drug therapy (prior antitumor treatment lines ≤4 lines) : relapse and/or refractory.
  2. Availability of qualified tissue samples by patient for pathological diagnosis by the central laboratory.
  3. The Eastern cooperative oncology group (ECOG) score 0-1.
  4. Life expectancy ≥ 3 months before starting HH2853 treatment.
  5. Sufficient bone marrow, liver and renal functions.

Exclusion Criteria:

* main criteria:

  1. Previous treatment with EZH2 or EZH1/2 inhibitors.
  2. Central nervous system invasion.
  3. Any previous history of bone marrow malignancy, including myelodysplastic syndrome (MDS).
  4. Received medications that are known potent CYP3A4 inducers/inhibitors within 1 week prior to first dose.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2022-07-27 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Phase Ib: To determine the RP2D of HH2853 in PTCL patients | 28-day treatment cycles
  Determine RP2D of HH2853
Phase II: To evaluate the efficacy of HH2853 of R/R PTCL patients who have received at least one prior systemic combination chemotherapy and at least one new drug | 28-day treatment cycles
  ORR will be based on the blinded independent review committee (BIRC). Assessment of oncologic response will be performed according to the 2014 edition of the Lugano Criteria for Efficacy [Lugano]

SECONDARY OUTCOMES:
Phase Ib: 1. Preliminary efficacy of HH2853 in R/R PTCL patients; | 28-day treatment cycles
  Investigator assessed: complete response rate (CRR)
Phase Ib: 1. Preliminary efficacy of HH2853 in R/R PTCL patients; | 28-day treatment cycles
  Duration of response (DoR)
Phase Ib: 1. Preliminary efficacy of HH2853 in R/R PTCL patients; | 28-day treatment cycles
  Disease control rate (DCR)
Phase Ib: 1. Preliminary efficacy of HH2853 in R/R PTCL patients; | 28-day treatment cycles
  Time to response (TTR)
Phase Ib: 2.To characterize the pharmacokinetic profile of HH2853 | 28-day treatment cycles
  Area under the concentration-time curve (AUC)
Phase Ib: 2.To characterize the pharmacokinetic profile of HH2853 | 28-day treatment cycles
  Maximum plasma concentration (Cmax)
Phase Ib: 2.To characterize the pharmacokinetic profile of HH2853 | 28-day treatment cycles
  Trough concentration (Cmin)
Phase Ib: 2.To characterize the pharmacokinetic profile of HH2853 | 28-day treatment cycles
  Time to maximum plasma concentration (Tmax)
Phase Ib: 2.To characterize the pharmacokinetic profile of HH2853 | 28-day treatment cycles
  Apparent clearance (CL/F)
Phase Ib: 2.To characterize the pharmacokinetic profile of HH2853 | 28-day treatment cycles
  Terminal half-life (t1/2)
Phase II: 1.To further assess the other efficacy of HH2853 of R/R PTCL patients who have received at least one prior systemic combination chemotherapy and at least one new drug (such as Chidamide, Pralatrexate and Brentuximab vedotin, et al.) therapy | 28-day treatment cycles
  ORR assessed by investigator
Phase II: 1.To further assess the other efficacy of HH2853 of R/R PTCL patients who have received at least one prior systemic combination chemotherapy and at least one new drug (such as Chidamide, Pralatrexate and Brentuximab vedotin, et al.) therapy | 28-day treatment cycles
  Complete response rate (CRR)
Phase II: 1.To further assess the other efficacy of HH2853 of R/R PTCL patients who have received at least one prior systemic combination chemotherapy and at least one new drug (such as Chidamide, Pralatrexate and Brentuximab vedotin, et al.) therapy | 28-day treatment cycles
  Progression-free survival (PFS)
Phase II: 1.To further assess the other efficacy of HH2853 of R/R PTCL patients who have received at least one prior systemic combination chemotherapy and at least one new drug (such as Chidamide, Pralatrexate and Brentuximab vedotin, et al.) therapy | 28-day treatment cycles
  Duration of response (DoR)
Phase II: 1.To further assess the other efficacy of HH2853 of R/R PTCL patients who have received at least one prior systemic combination chemotherapy and at least one new drug (such as Chidamide, Pralatrexate and Brentuximab vedotin, et al.) therapy | 28-day treatment cycles
  Disease control rate (DCR)
Phase II: 1.To further assess the other efficacy of HH2853 of R/R PTCL patients who have received at least one prior systemic combination chemotherapy and at least one new drug (such as Chidamide, Pralatrexate and Brentuximab vedotin, et al.) therapy | 28-day treatment cycles
  Time to response (TTR)
Phase II: 1.To further assess the other efficacy of HH2853 of R/R PTCL patients who have received at least one prior systemic combination chemotherapy and at least one new drug (such as Chidamide, Pralatrexate and Brentuximab vedotin, et al.) therapy | 28-day treatment cycles
  Overall survival (OS) by BIRC
Phase II: 1.To further assess the other efficacy of HH2853 of R/R PTCL patients who have received at least one prior systemic combination chemotherapy and at least one new drug (such as Chidamide, Pralatrexate and Brentuximab vedotin, et al.) therapy | 28-day treatment cycles
  Overall survival (OS) by investigator
Phase II: 2. To evaluate the safety and tolerability of HH2853 | 28-day treatment cycles
  Duration and severity of adverse events (AEs)
Phase II: 3. To characterize the population pharmacokinetic profile of HH2853 | 28-day treatment cycles
  Area under the concentration-time curve (AUC)
Phase II: 3. To characterize the population pharmacokinetic profile of HH2853 | 28-day treatment cycles
  Maximum plasma concentration (Cmax)
Phase II: 3. To characterize the population pharmacokinetic profile of HH2853 | 28-day treatment cycles
  Steady-state trough concentration (Cmin)
Phase II: 3. To characterize the population pharmacokinetic profile of HH2853 | 28-day treatment cycles
  Time to maximum plasma concentration (Tmax)
Phase II: 3. To characterize the population pharmacokinetic profile of HH2853 | 28-day treatment cycles
  Apparent clearance (CL/F)
Phase II: 3. To characterize the population pharmacokinetic profile of HH2853 | 28-day treatment cycles
  Half life (t1/2)

OTHER OUTCOMES:
Phase Ib and II: 1. To explore biomarkers related to response and effect of HH2853 | 28-day treatment cycles
  mutation status of EZH2
Phase Ib and II: 2. To explore the correlation between HH2853 exposure with safety, efficacy and pharmacokinetic parameters | 28-day treatment cycles
  Correlation between exposure (Cmax or AUC) and safety/efficacy/pharmacodynamic biomarkers (trimethylation of histone H3 at lysine 27 [H3K27me3])

CONTACTS AND LOCATIONS:
Overall Officials: Tongyu Li, MD, Principal Investigator — Sichuan Cancer Hospital and Research Institute
Locations (1):
- Sichuan Cancer Hospital, Chengdu, Chengdu, China

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD based on business strategy.